CLINICAL TRIAL: NCT00086970
Title: A Phase I Study Of BG In Combination With Ifosfamide For Advanced Solid Tumors
Brief Title: Ifosfamide With or Without O(6)-Benzylguanine in Treating Patients With Unresectable, Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02601; 12999B; U01CA069852 (NIH); CDR0000371909 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Ifosfamide; indolepropanol phosphate; O(6)-benzylguanine

ARMS (2):
- Arm I (ifosfamide) (Experimental): Patients receive high-dose ifosfamide IV continuously over 72 hours on days 1-3.
  Interventions: Drug: ifosfamide
- Arm II (O6-benzylguanine, ifosfamide) (Experimental): Patients receive a bolus dose of O6-benzylguanine (BG) IV over 1 hour on day 1 followed by BG IV continuously and high-dose ifosfamide IV continuously over 72 hours on days 1-3.
  Interventions: Drug: ifosfamide; Drug: O6-benzylguanine

INTERVENTIONS:
Drug: ifosfamide — Given IV
  Other Names: Cyfos; Holoxan; IFF; IFX; IPP
Drug: O6-benzylguanine — Given IV
  Other Names: BG
  Arms: Arm II (O6-benzylguanine, ifosfamide)

SUMMARY:
This randomized phase I trial is studying the side effects and best dose of O(6)-benzylguanine when given together with ifosfamide and to see how well it works compared to ifosfamide alone in treating patients with unresectable metastatic solid tumors. Drugs used in chemotherapy, such as ifosfamide and O(6)-benzylguanine, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining ifosfamide with O(6)-benzylguanine may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of O6-benzylguanine when administered with standard high-dose ifosfamide in patients with unresectable, metastatic solid tumors.

II. Determine whether O6-benzylguanine enhances ifosfamide-mediated myelosuppression in patients treated with this regimen.

III. Determine the relationship between O6-benzylguanine dose and intra-individual variability in the degree of myelosuppression in patients treated with this regimen.

IV. Determine the safety and toxicity of this regimen in these patients.

SECONDARY OBJECTIVES:

I. Determine the effect of O6-benzylguanine on pharmacodynamic endpoints, including apoptosis and DNA damage, in patients treated with this regimen.

II. Determine the pharmacokinetics of O6-benzylguanine and its major metabolite, 8-oxoBG, in patients treated with this regimen.

OUTLINE: This is a randomized, open-label, multicenter, dose-escalation study of O6-benzylguanine.

Course 1: All patients receive high-dose ifosfamide IV continuously over 72 hours on days 1-3.

Course 2: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive high-dose ifosfamide as in course 1.

Arm II: Patients receive a bolus dose of O6-benzylguanine (BG) IV over 1 hour on day 1 followed by BG IV continuously and high-dose ifosfamide IV continuously over 72 hours on days 1-3. Cohorts of 6-12 patients receive escalating doses of BG (administered as a bolus and as a continuous infusion during course 2) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 6 or 4 of 12 patients experience dose-limiting toxicity.

Course 3 and all subsequent courses: All patients receive BG (at the MTD determined in course 2, arm II) and high-dose ifosfamide as in course 2, arm II. In all courses, all patients also receive filgrastim (G-CSF) beginning on day 5 and continuing until blood counts recover. In all courses and in both arms, treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor

  * Unresectable, metastatic disease
  * No primary tumors
* Eligible for high-dose ifosfamide-based therapy
* No known brain metastases
* Performance status - ECOG 0-1
* Performance status - Karnofsky 70-100%
* More than 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* AST and ALT ≤ 2.5 times upper limit of normal
* Bilirubin normal
* Creatinine normal
* Creatinine clearance ≥ 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to O6-benzylguanine or other study agents
* No concurrent uncontrolled illness
* No active or ongoing infection
* No psychiatric illness or social situation that would preclude study compliance
* More than 24 hours since prior colony-stimulating factors (filgrastim [G-CSF] or sargramostim [GM-CSF])
* No prior hematopoietic stem cell transplantation
* No concurrent pegfilgrastim
* No concurrent immunotherapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No other concurrent chemotherapy
* No concurrent hormonal therapy
* More than 4 weeks since prior radiotherapy and recovered
* No concurrent therapeutic radiotherapy
* More than 4 weeks since prior anticancer therapy
* No more than 2 prior cytotoxic regimens
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer agents or therapies
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-06; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Change in degree of myelosuppression (thrombocytopenia and neutropenia) quantified by both duration of neutropenia and severity of neutropenia | Baseline up to 1 year
Maximum tolerated dose (MTD) of O6-benzylguanine defined as the dose preceding that at which 3 of 6 or 4 of 12 patients experience dose-limiting toxicity | 21 days
  DLT is defined as any >= grade 3 non-hematologic toxicity, grade 4 thrombocytopenia, or prolonged neutropenia.

SECONDARY OUTCOMES:
Pharmacodynamics including apoptosis and DNA damage | Up to 1 year
Pharmacokinetics of O6-benzylguanine | Up to day 3 of course 2
  Summarized using descriptive statistics (mean, median, standard deviation, and interquartile range). Estimated via nonlinear regression.

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Smith, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States